CLINICAL TRIAL: NCT04889768
Title: HIPEC Combined With Camrelizumab, Paclitaxel and S-1 for Conversion Therapy in Patients With Advanced Gastric Cancer With Peritoneal Metastasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2021-63
Record Dates: First submitted 2021-05-12; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-03

CONDITIONS: Gastric Cancer, HIPEC, Anti-PD-1 Antibody Camrelizumab (SHR-1210), Chemotherapy and Surgery
MeSH Terms: conditions — Stomach Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy; camrelizumab; Drug Therapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: HIPEC, anti-PD-1 antibody Camrelizumab (SHR-1210), Chemotherapy and Surgery (Experimental): 1. surgical exploration, if PCI<20, then we perform this study.
  2. HIPEC: Taxol (Paclitaxel Injection) 75 mg/m2, d1, d3 within 72 hours after surgical exploration; oral chemotherapy:S-1: 80mg/m2, twice daily for d1-d14, and then suspend for one week; Intravenous drip anti-PD-1 antibody Camrelizumab (SHR-1210) 200mg fixed dose every 3 weeks.
  3. Chemotherapy and PD-1 treatment (4 cycles) : Taxol 150mg/m2,d1; S-1: 80-120mg/m2, twice daily for two weeks, and then suspend for one week; Camrelizumab (SHR-1210) 200mg fixed dose every 3 weeks.
  4. Surgery: Secondary surgical exploration: if PCI less than 20, then assess the patient's condition and consider whether perform the cytoreductive surgery (resection of primary tumors and metastases ). For inoperable patients, continue to use this program for treatment.
  5. After the surgery, HIPEC for two cycles, anti-PD-1 antibody Camrelizumab (SHR-1210) for 4 cycles, and PS chemotherapy for 4 cycles.
  Interventions: Drug: HIPEC, anti-PD-1 antibody Camrelizumab (SHR-1210), Chemotherapy and Surgery

INTERVENTIONS:
Drug: HIPEC, anti-PD-1 antibody Camrelizumab (SHR-1210), Chemotherapy and Surgery — 1. HIPEC: Taxol (Paclitaxel Injection) 75 mg/m2, d1, d3 within 72 hours after surgical exploration; oral chemotherapy:S-1: 80mg/m2, twice daily for d1-d14, and then suspend for one week; Intravenous drip anti-PD-1 antibody Camrelizumab (SHR-1210) 200mg fixed dose every 3 weeks.
  2. Chemotherapy and PD-1 treatment (4 cycles) : Taxol 150mg/m2,d1; S-1: 80-120mg/m2, twice daily for two weeks, and then suspend for one week; Camrelizumab (SHR-1210) 200mg fixed dose every 3 weeks.
  3. Surgery: Secondary surgical exploration: if PCI less than 20, then assess the patient's condition and consider whether perform the cytoreductive surgery (resection of primary tumors and metastases ). For inoperable patients, continue to use this program for treatment.
  4. After the surgery, HIPEC for two cycles, anti-PD-1 antibody Camrelizumab (SHR-1210) for 4 cycles, and PS chemotherapy for 4 cycles.

SUMMARY:
There is no currently available treatment for peritoneal metastasis of gastric cancer. Hyperthermic intraperitoneal chemotherapy (HIPEC) can not only maintain the high concentration of drugs in the abdominal cavity, but also improve the anti-tumor efficacy of chemotherapy drugs through the thermo-thermal effect. In recent years, immunotherapy has made great progress in the treatment of gastric cancer. We want to explore the hyperthermic intraperitoneal chemotherapy (HIPEC) combined with Camrelizumab (SHR-1210) and intravenous chemotherapy for Creating the Operation Chance in advanced gastric cancer with peritoneal metastasis.

DETAILED DESCRIPTION:
To assess the effectiveness and safety of Hyperthermic intraperitoneal chemotherapy, anti-PD-1 antibody Camrelizumab (SHR-1210), intravenous chemotherapy combined with surgery for the treatment of advanced gastric cancer with peritoneal metastasis, so as to further find out the optimal protocol for the Conversion therapy in the patients with advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced gastric (gastroesophageal junction) adenocarcinoma confirmed by histology/cytology and negative for HER-2 by IHC/FISH
2. The presence of gastric cancer peritoneal metastasis is confirmed by laparoscopic exploration, and the PCI≤20
3. Untreated (e.g. radiotherapy, chemotherapy, target therapy and immunotherapy)
4. ECOG (Eastern Cooperative Oncology Group) : 0~1
5. There is at least one measurable lesion according to the RECISTv1.1
6. Normal hemodynamic indices before the recruitment
7. Good cardiac function before the recruitment, no seizure of myocardial infarction in past half year, and controllable hypertension and other coronary heart diseases
8. Fertile female subjects must undergo a serum-negative pregnancy test within 72 hours before starting the study drug and must agree to use a medically approved effective contraceptive during the study period and within 180 days of the last dose of the study drug; Male subjects whose partners are women of child-bearing age should undergo surgical sterilization or agree to use effective methods of contraception during the study period and within 180 days of the last study administration.
9. Signed the Informed Consent Form

Exclusion Criteria:

1. Immunosuppressive drugs were used within 30 days before the first use of carrlizumab, excluding nasal spray and inhaled corticosteroids or systemic steroids in physiological dose (i.e. no more than 10 mg / day of prednisolone or other corticosteroids in physiological dose of the same drug)
2. There is any active autoimmune disease or a history of autoimmune disease (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism; subjects with vitiligo or asthma in childhood have been completely relieved, and those who do not need any intervention after adulthood can be included Asthma requiring medical intervention with bronchodilator was not included.) Distal metastasis to lung, liver, or paraaortic lymph node metastasis
3. Ever operation on the stomach
4. Serious diseases that are difficult to control
5. Allergy to the drugs in this protocol
6. There are many factors that affect the absorption of oral drugs, including inability to swallow, chronic diarrhea, intestinal obstruction and so on.
7. The peripheral neuropathy was more than 1 grade
8. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), active hepatitis B (HBV DNA ≥ 500 IU / ml), hepatitis C (HCV antibody positive, and HCV RNA higher than the detection limit of the analysis method) or co infection with hepatitis B and C.
9. Active infection (e.g. intravenous drip of antibiotics, antifungal or antiviral drugs) or fever of unknown origin >38.5℃ 1 weeks ago (except for tumor related fever determined by researchers).
10. Abnormal coagulation (INR > 1.5 or APTT > 1.5 × ULN), bleeding tendency or undergoing thrombolysis or anticoagulation. Long term anticoagulation with warfarin or heparin or long-term antiplatelet therapy is required.
11. The live attenuated vaccine shall be inoculated within 4 weeks before the first administration or during the study period
12. Any other malignant tumor has been diagnosed within 3 years before the study, except for basal cell or squamous cell skin cancer or cervical carcinoma in situ which has been fully treated
13. A history of psychoactive substance abuse or abuse is known
14. The presence of other serious physical or mental illness or laboratory abnormalities may increase the risk of participating in the study, or interfere with the results of the study, as well as the patients who the investigator believes are not suitable for participating in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-07-31 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
R0 resection | 3 months
  the rate of R0 resection

SECONDARY OUTCOMES:
Overall survival time | 3 years
  the overall survival time
Disease-Free Survival | 3 years
  Disease-Free Survival of participants with with advanced gastric cancer with peritoneal metastasis followed by surgery
ORR | 3 years
  Objective Response Rate
Adverse Events | 3 years
  Number and degree of Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- The Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital), Hangzhou, China